CLINICAL TRIAL: NCT05942547
Title: Clinical Study Evaluating the Efficacy and Safety of Diosmin on Non-diabetic Patients With Non-alcoholic Steatohepatitis.
Brief Title: the Efficacy and Safety of Diosmin on Non-diabetic Patients With Non-alcoholic Steatohepatitis.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Merna Tarek Elsaeed, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3626MS202/6/23
Record Dates: First submitted 2023-06-21; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diosmin

STUDY DESIGN:
Intervention Model Description: This study will be a randomized double-blind placebo-controlled parallel study that will involve 48 non-diabetic patients with confirmed diagnosis of NASH.
  . The patients will be randomized in a 1:1 ratio by a neutral researcher using sealed envelopes methods with assignment codes for each available allocation to receive either diosmin 600 mg twice daily (Diosmin group; n = 24) or placebo twice daily (Placebo group; n = 24). The study duration will be 12 weeks.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diosmin group (Experimental): (Diosmin group; n = 24):will receive 600 mg twice daily
  Interventions: Drug: Diosmin
- placebo group (Placebo Comparator): placebo group n=24 :will receive placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diosmin — diosmin 600mg twice daily
  Arms: diosmin group
Drug: Placebo — twice daily
  Arms: placebo group

SUMMARY:
This is a randomized, controlled study evaluating diosmin tablets administered daily for 3 months. The purpose of the study is to evaluate the efficacy and safety of diosmin on non-diabetic patients with non-alcoholic steatohepatitis.

DETAILED DESCRIPTION:
The aim of the study is to test the implication of diosmin in fatty liver disease through evaluation of its efficacy and safety in non-diabetic patients with nonalcoholic steatohepatitis (NASH).

Patients and Methods:

This study will be a randomized double-blind placebo-controlled parallel study that will involve 48 non-diabetic patients with confirmed diagnosis of NASH. The patients will be recruited from outpatient Clinic of the internal medicine department, Tanta University Hospital, Tanta, Egypt. The diagnosis of NASH will be confirmed by imaging technique (increased liver echogenicity, stronger echoes in the hepatic parenchyma, vessel blurring, and narrowing of the lumen of the hepatic veins), mild to moderate elevation in aminotransferase activities (>2 but <5 times upper limit of normal), hepatic steatosis index (HIS) >36, HAIR score (hypertension, alanine aminotransferase level, insulin resistance) of 2 or 3 and cytokeratin-18 level >240 IU/L. The patients will be randomized in a 1:1 ratio by a neutral researcher using sealed envelopes methods with assignment codes for each available allocation to receive either diosmin 600 mg twice daily (Diosmin group; n = 24) or placebo twice daily (Placebo group; n = 24). The study duration will be 12 weeks.

* All participants and will be informed about the benefits and risks of the study. The expected risks that will be clarified to patients include diosmin related adverse effect; stomach pain, diarrhea, headache, skin redness, muscle pain, and altered heart rate.
* Any unexpected risks that will appear during the course of the research will be clarified to the participants and to the ethical committee on time. The data of the enrolled patients will be confidential.
* All enrolled patients will give their written informed consents. The study will be carried out between june2023 and june2025.Demography and anthropometric measurements At baseline and after intervention, all participants will be submitted to medical history taking, demography (age, sex, and medication history), physical examination with heart rate evaluation, measurement of weight and height with subsequent calculation of body mass index (BMI)=[Weight (kg)÷ Height2 (m)]. 2. Ultrasonographic examination Ultrasonography of the liver will be carried out at baseline and at the end of the study by the same operator. Ultrasonography Fatty Liver Indicator (US-FLI) is a scoring system ranging 2-8 based on the intensity of liver/kidney contrast, posterior attenuation of ultrasound beam, vessel blurring, difficult visualization of gallbladder wall, and difficult visualization of the diaphragm and areas of focal sparing. NAFLD is diagnosed by the minimum score ≥2. 3. Blood samples collection and biochemical measurements Before and after the intervention, 8 ml of venous blood will be withdrawn by antecubital venipuncture from each participant after overnight fasting (12 h fasting period) between 8:30 and 10:30 a.m. into plain test tubes. Three ml of the blood samples will be used for the assessment of complete blood count. The remaining 5 ml of blood will be centrifuged at 3000 rpm for 10 min. The separated serum will be divided into two portions. The first portion will be used for immediate determination of liver panel, fasting lipid profile and fasting blood glucose concentration. The second portion of the serum will be frozen at-80°C until analysis of the remaining parameters including malondialdehyde (MDA), tumor necrosis factor- alpha (TNF-α), fasting insulin and transforming growth factor-beta1 (TGF-β1).
* Complete blood count (CBC) will be determined by automated hematology analyzer.
* Liver enzymes (AST, ALT, and GGT) will be determined by kinetic method.
* Serum albumin level which will be assayed by colorimetric bromocresol green method or other available method.
* Fasting blood glucose will be determined by glucose oxidase method or glycated hemoglobin (HbA1c%) will be measured by commercially available method
* Lipid panel including total cholesterol (TC), triglyceride (TG) and HDLC will be assessed by enzymatic colorimetric method.
* Fasting insulin level will be determined by ELISA.
* Malondialdehyde (MDA) which will be assessed by colorimetric method.
* Tumor necrosis factor- alpha (TNF-α) will be determined by ELISA.
* Serum transforming growth factor-beta1 (TGF-β1) will be determined by ELISA.
* In addition, prothrombin time (PT) or INR will be assessed regularly at baseline and on monthly basis. 4. Calculated parameters
* Low density lipoprotein cholesterol (LDL-C) will be calculated using the

Friedewald formula17 as follows:

* [LDL-C=TC- HDL-C- (TG÷5)] provided that TG level is less than 400 mg/dl.

  * Very low density lipoprotein cholesterol will be calculated using the Friedewald formula17 as follows: o VLDL = TG/5.
  * The Homeostasis Model Assessment-insulin resistance (HOMA-IR) 18 will be calculated as follow: o HOMA-IR= (Fasting glucose × fasting insulin/405) when glucose is expressed by mg/dl and insulin is expressed by μIU/ml.
  * Hepatic steatosis index "HSI".
* Hepatic steatosis index includes gender, history of type 2 diabetes mellitus (T2DM), BMI, alanine transaminase "ALT", and aspartate transaminase "AST".
* HSI is calculated by the following formula:

  8 × (ALT/AST ratio) + BMI + 2 if female and + 2 if diabetic (0 since the study will be conducted on non-diabetic).
* HAIR score "hypertension, alanine aminotransferase level, insulin resistance". It is calculated from hypertension ≥140/90, ALT >40 and HOMA-IR >5.
* Presence of one item indicates HAIR score=1. o Presence of two item indicates HAIR score=2.
* Prescience of the 3 items indicates HAIR score=3.

  - Fibrosis risk scores: o Fibrosis index based on the 4 factors (FIB-4). FIB-4= Age (years) × AST (IU/l)/[platelet count (109

  /L) ×√ ALT (IU/l)].
* Aspartate transaminase-to-platelet ratio index (APRI).22 APRI =AST (IU/l)/(upper limit of normal) X 100 /platelet count (109

  /L).
* NAFLD fibrosis score (NFS) which depends on 7 parameters including age, BMI, diabetes, AST, ALT, platelets count, and albumin concentration.

  * Score <-1.455 predicts absence of significant fibrosis (F0-F2).
  * Score ≤ - 1.455- ≤ 0.675 predicts intermediate score
  * Score > 0.675 predicts presence of significant fibrosis (F3-F4).

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic patients with or without hypertension.
* Both males and females.
* Age >18 years old.
* Overweight and obese patient: Body mass index (BMI) ≥ 25 kg/m2 <.40 kg/m2
* Patients with established diagnosis of NASH based on liver ultrasonography, mild to moderate elevation in aminotransferase activities (>2 but <5 times upper limit of normal), hepatic steatosis index (HIS) >36, HAIR score of 2 or 3.

Exclusion Criteria:

* Patients with BMI ≥ 40 kg/m2
* Patients with type 2 diabetes mellitus (T2DM) on the basis of a fasting plasma glucose (FPG) level ≥ 126 mg/dl (7mmol/L) or glycated hemoglobin (HbA1c) > 6.5% (48 mmol/mol).
* Alcohol consumption greater than 20 g per day for women or greater than 30 g for men for at least three consecutive months over the past 5 years.
* History of viral hepatitis, hemochromatosis, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis, sclerosing cholangitis, biliary obstruction, alpha-1 antitrypsin deficiency.
* Patients on medications interfere with lipid and carbohydrate metabolism (statin, fibrate, beta blockers, thiazide, corticosteroids, etc).
* Patients with cancer or with a history of cancer.
* Patients with thyroid disorder.
* Patients on medications associated with steatosis such as NSAIDs, amiodarone, tamoxifen, estrogen, sodium valproate, corticosteroids, and methotrexate.
* Patients with inflammatory diseases (rheumatoid arthritis, ulcerative colitis, etc).
* Patients on supplements known to have antioxidant activity such as vitamin E, vitamin C, zinc, and selenium.
* Patient with a history of cardiovascular diseases.
* Patients with arrhythmia or altered heart rate.
* Patients on blood thinning agents (warfarin, clopidogril, aspirin, etc), anticonvulsants (carbamazepine and phenytoin), muscle relaxants (chlorzoxazone) and non-steroidal anti-inflammatory drugs (diclofenac( in order to avoid potential pharmacodynamics and pharmacokinetic drug interactions with diosmin.
* Pregnant and breastfeeding women.
* Females on oral contraceptive pills will be also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-10 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
the change in ultrasound including NAFLD fibrosis scor | at baseline then after 3 months
  The change in ultrasound through decreasing liver echogenicity, Lower echoes in the hepatic parenchyma, no vessel blurring, and decrease narrowing of the lumen of the hepatic veins Ultrasonography Fatty Liver Indicator (US-FLI) <2
The change in fibrosis risk score | at baseline then after 3 months
  Score <-1.455 predicts absence of significant fibrosis (F0-F2)

SECONDARY OUTCOMES:
The secondary outcome is the change in biological biomarkers and other measured parameters | at baseline then after 3 months
  The change in liver panel
secondary outcome is the change in biological biomarkers and other measured parameters | at baseline then after 3 months
  The change in the Homeostasis Model Assessment-insulin resistance (HOMA-IR)
secondary outcome is the change in biological biomarkers and other measured parameters | at baseline then after 3 months
  The change in biological parameters (MDA, TNF-α, and TGF-β1)

CONTACTS AND LOCATIONS:
Overall Officials: tarek mohamed mostafa, professor, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No